CLINICAL TRIAL: NCT02531152
Title: A Randomized, Observer-masked Study of the Safety, Tolerability and Pharmacodynamics of Sequential Ascending 28-Day Repeated Topical Doses of SAR366234 Versus Latanoprost in Patients With Open Angle Glaucoma or Ocular Hypertension
Brief Title: 28-Day Repeated Topical Study to Evaluate the Safety and Activity of 5 Escalating Dose Levels of SAR366234 and One Dose of Latanoprost in Patients With Open Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TDR13459; U1111-1153-3544 (Other: UTN)
Record Dates: First submitted 2015-08-20; First posted 2015-08-24 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Open Angle Glaucoma -Ocular Hypertension
MeSH Terms: interventions — Latanoprost

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- SAR366234 (Dose 1) (Experimental): A low dose of SAR366234 will be administered 2 drops per eye per day for 28 days
  Interventions: Drug: SAR366234
- SAR366234 (Dose 2) (Experimental): A medium dose of SAR366234 will be administered 1 drop per eye per day for 28 days
  Interventions: Drug: SAR366234
- SAR366234 (Dose 3) (Experimental): A medium dose of SAR366234 will be administered 2 drops per eye per day for 28 days
  Interventions: Drug: SAR366234
- SAR366234 (Dose 4) (Experimental): A high dose of SAR366234 will be administered 1 drop per eye per day for 28 days
  Interventions: Drug: SAR366234
- SAR366234 (Dose 5) (Experimental): A high dose of SAR366234 will be administered 2 drops per eye per day for 28 days
  Interventions: Drug: SAR366234
- Latanoprost (Active Comparator): A dose of Latanoprost will be administered 1 drop per eye per day for 28 days
  Interventions: Drug: Latanoprost

INTERVENTIONS:
Drug: Latanoprost
  Other Names: Xalatan
  Arms: Latanoprost
Drug: SAR366234
  Arms: SAR366234 (Dose 1); SAR366234 (Dose 2); SAR366234 (Dose 3); SAR366234 (Dose 4); SAR366234 (Dose 5)

SUMMARY:
Primary Objective:

To assess the local and systemic safety and tolerability of ascending repeated topical doses of SAR366234 monotherapy in patients with open angle glaucoma (OAG) or ocular hypertension (OHT) as compared to latanoprost.

Secondary Objective:

To assess the pharmacodynamic activity of ascending repeated topical doses of SAR366234 in patients with OAG or OHT as compared to latanoprost.

DETAILED DESCRIPTION:
The total study duration for one patient is up to 11 weeks, including a screening period of up to 6 weeks run-in (depending on washout requirements), a 4-week treatment period, and a 1-week follow-up period.

The study design is also a parallel cohort study to assess the safety, tolerability, and pharmacodynamic activity of SAR366234.

ELIGIBILITY:
Inclusion criteria:

* Male or female patients ≥18 years of age.
* Patients diagnosed with OAG (including pseudoexfoliation and pigment dispersion syndromes and patients with a history of narrow angle closure with a patent peripheral iridotomy) or OHT.
* Documented intraocular pressure (IOP) fulfilling the eligibility criteria (below) at both the screening and baseline visits:
* At the screening visit
* an IOP ≤21 mmHg in both eyes if currently treated with an IOP-lowering medication or
* an IOP ≥22 mmHg and <36 mmHg if treatment-naïve or not on IOP lowering medication for at least 5 weeks.
* At the baseline visit following washout
* an IOP ≥22 mmHg and <36 mmHg at about 8:00 am,
* an IOP >20 mmHg and <36 mmHg at about 12:00 noon, and
* an IOP >18 mmHg and <36 mmHg at about 4:00 pm.
* Baseline laboratory parameters within the defined screening threshold for the Investigator site, unless the Investigator considers and documents an abnormality to be clinically irrelevant.
* Having given written informed consent prior to undertaking any study-related procedure, including stopping their current glaucoma treatment, if any, and engaging into the corresponding washout procedures.
* Patients should agree to discontinue any concomitant topical ocular medication(s) and current IOP-reducing agents.
* Best corrected Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity score of +1.0 logMAR (Snellen equivalent 20/200) or better in both eyes at the screening and baseline visits.
* Patients on systemic β blockers must be on a stable dose for at least 2 weeks before screening and should expect to continue the treatment during the study with no anticipated alteration in the medication dose.
* Patients should agree to discontinue contact lenses during treatment with the study medication.

Exclusion criteria:

* Any clinically significant disease or concomitant medication that would interfere with the study evaluation.
* Patients with advanced glaucoma at risk of progression during the study in the opinion of the Investigator.
* Presence or history of hypersensitivity to latanoprost or known history of non-response to any prostaglandin analog given for the reduction of IOP.
* History of hypersensitivity or allergy to any component of the investigational medicinal product or any of the diagnostic medications or materials used in the conduct of the study.
* Use or expected need for ocular (topical, periocular, or intravitreal), local (inhaled or nasal), or systemic glucocorticoid medications within 4 weeks prior to the baseline visit and for the duration of the study.
* Any vaccination within the last 28 days from randomization or during screening whichever is longer.
* Any patient in the exclusion period of a previous study according to applicable regulations.
* Any patient who cannot be contacted in case of emergency.
* Any patient who is the Investigator or any subinvestigator, research assistant, pharmacist, study coordinator, or other staff thereof, directly involved in conducting the study.
* Positive result on any of the following tests: hepatitis B surface (HBs Ag) antigen, anti-hepatitis C virus (anti-HCV) antibodies, anti-human immunodeficiency virus 1 and 2 antibodies (anti-HIV1 and anti HIV2 Ab).
* Positive result on urine drug screen (amphetamines/methamphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, opiates) unless the result of a medical prescription.
* An IOP ≥36 mmHg at any time during the screening, baseline, or randomization visits (Day 1 predose).
* History of ocular surgery (including laser) or trauma in either eye within 6 months of the screening visit.
* History of glaucoma filtering surgery or aqueous shunt procedures (traditional valves and/or microinvasive glaucoma surgery [MIGs]).
* History of ocular infection within the past 3 months or ongoing or recurrent ocular inflammation (ie, moderate to severe blepharitis, allergic conjunctivitis, herpetic keratitis, peripheral ulcerative keratitis, scleritis, or uveitis) in either eye. Any ocular abnormalities or symptoms indicative of ongoing ophthalmic disease (except if related to glaucoma or OHT).
* Central corneal thickness <500 µm or >620 µm at the baseline visit.
* Any evidence of cornea guttata or corneal endothelial dysfunction from medical history or at the baseline visit.
* Uncontrolled disease that would interfere with the study conduct, the interpretation of the study results, or the ability of the patient to meet the requirements of the study schedule.
* Any corneal abnormalities preventing reliable applanation tonometry.
* Closed/barely open anterior chamber angle or a history of acute angle closure in either eye not adequately treated with a peripheral iridectomy.
* Diagnosis of a clinically significant or progressive retinal disease (eg, diabetic retinopathy, advanced age-related macular degeneration, inherited retinal dystrophies) in either eye.
* Advanced optic nerve abnormality or history of visual field loss in either eye based on the assessment of the Investigator which could put the patient at risk of glaucoma progression by participating in the study.
* History of aphakia, pseudophakia with a torn posterior lens capsule, macular edema, or known risk factors for macular edema in either eye.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Number of adverse events (including local tolerance and ophthalmological examinations) | From screening (Day -42) up to approximately Day 39

SECONDARY OUTCOMES:
Assessment of IOP using Goldman applanation tonometry | From screening (Day -42) up to approximately Day 39

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (5):
- United States (5):
  - Investigational Site Number 840001, Inglewood, California
  - Investigational Site Number 840003, Cape Coral, Florida
  - Investigational Site Number 840005, Roswell, Georgia
  - Investigational Site Number 840004, Saint Joseph, Michigan
  - Investigational Site Number 840002, Memphis, Tennessee